CLINICAL TRIAL: NCT05268679
Title: Study of the Humoral and Cellular Response to Vaccines Against SARS-CoV-2 in Heart Transplant Recipients
Brief Title: Covid-19 Vaccine Response in Heart Transplant Recipients
Acronym: COVHEART
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211456
Record Dates: First submitted 2022-03-04; First posted 2022-03-07 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Heart Transplantation; COVID-19 Virus Infection; COVID-19 Vaccine
Keywords: Heart transplant recipients; Covid-19 virus infection; SARS-CoV-2 vaccine; Vaccine Effectiveness; Humoral immune response; Cellular Immune Response
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart transplant recipients: Heart transplant recipients followed at Bichat Hospital and who were offered vaccination against SARS-CoV-2, regardless of whether they agreed to be vaccinated or not.
  Interventions: Other: Biospecimen Collection; Other: Questionnaire; Other: Electronic Health Record Review

INTERVENTIONS:
Other: Biospecimen Collection — A blood of a sample of 2 x 7 mL will be collected for the analysis of the anti-SARS-CoV-2 T-cell response during a scheduled check-up as part of their routine follow-up
Other: Questionnaire — Patients who have received SARS-CoV-2 vaccination will be asked to complete the Vaccine tolerance questionnaire
Other: Electronic Health Record Review — For heart transplant recipients who were offered vaccination against SARS-CoV-2 medical records will be reviewed retrospectively.

SUMMARY:
Clinical studies indicate a decrease in vaccine efficacy in certain immunocompromised populations (kidney transplant recipients, patients undergoing chemotherapy). It was recently reported that only 18% to 49% of heart transplant recipients developed antibodies after 2 doses of BNT162b2 vaccine. Following the published results, it is currently recommended to use 3 doses in organ transplant recipients who have not contracted COVID-19 and 2 doses in those who have been infected. The effectiveness of this strategy is not yet sufficiently evaluated in heart transplant recipients. Moreover, the factors associated with the humoral and cellular response, the kinetics and durability of the humoral response, the occurrence of the cellular immune response and the tolerance of the vaccine are not well known in this population.

To provide answers to these different questions, we set ourselves the objective of evaluating the humoral and cellular response to messenger RNA (mRNA) vaccines in heart transplant recipients followed at Bichat Hospital.

DETAILED DESCRIPTION:
In order to evaluate the effectiveness and safety of currently adopted vaccination strategies in heart transplant recipients we intend to study the humoral and cellular responses to SARS-CoV-2 mRNA vaccines in heart transplant recipients followed at Bichat Hospital.

All heart transplant recipients followed at Bichat Hospital will be invited to participate in this research.

The vaccination schedule was 3 doses for the seronegative patients without documented infection, and 2 doses for patients who were seropositive or had a positive Reverse Transcriptase - Polymerase Chain Reaction (RT-PCR) test for SARS-CoV-2. Most patients were vaccinated at Bichat Hospital. Their vaccination schedule will be recovered. Some patients refused vaccination.

Since the beginning of 2020, the transplant patients have benefited from systematic serological tests and RT-PCR testing of nasopharyngeal swabs in the event of symptoms suggestive of SARS-CoV-2 infection as part of routine care. The results of these tests will be retrieved from medical records retrospectively in order to investigate the kinetics and durability of the humoral response. Demographic and clinical data will be collected to determine the factors associated with vaccine response.

In addition, a whole blood sample will be drawn at inclusion in order to evaluate cellular response. The patients will be also asked to answer a questionnaire regarding vaccine tolerance.

The effectiveness of vaccination program will be assessed after 6-month follow-up based on the occurrence of SARS-CoV-2 infection, unscheduled medical consultation or hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplant patients followed at Bichat Hospital
* Aged 18 or older
* Informed and having expressed their non-objection to participation in this research
* Able to give their agreement

Exclusion Criteria:

* Minors
* Heart transplant recipients who have expressed their opposition to their participation
* Legally protected adult
* Persons under the State Medical Assistance (AME)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart transplant recipients followed at Bichat Hospital and who were offered vaccination against SARS-CoV-2, regardless of whether they agreed to be vaccinated or not.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Anti-SARS-CoV-2 neutralizing antibody levels | Change from baseline to month 6
  Anti-SARS-CoV-2 neutralizing antibody levels over time, with quantification of immunoglobulin G (IgG) directed against the Receptor Binding Domain (RBD) of the Spike (S) protein
Efficacy of COVID-19 Vaccines against SARS-CoV-2 infection | Day 0
  Search for memory T lymphocytes specific to SARS-CoV-2 using an Elispot interferon γ test during the inclusion visit

SECONDARY OUTCOMES:
Efficacy of COVID-19 vaccines against SARS-CoV-2 infection | Month 6
  Proportion of vaccinated heart transplant recipients having had an infection documented by RT-PCR and a serious infection requiring hospitalisation
Safety of COVID-19 vaccines | Day 0
  Patients will be asked to complete the Vaccine tolerance questionnaire where they will asses and evaluate their symptoms. These will include Diffuse muscle pain (on a scale of 10)/ Headache (on a scale of 10)/ Digestive disorders/ Skin rash/ Pain at the injection site (on a scale of 10)/ Fever/ Fatigue/ Other. Lower scores for all symptoms would indicate a better tolerance.
Kinetics of the humoral response | Change from baseline to month 6
  Change in SARS-CoV-2 Antibody Concentrations following mRNA COVID-19 vaccine series

CONTACTS AND LOCATIONS:
Overall Officials: Richard DORENT, MD, Principal Investigator — AP-HP, Bichat-Claude Bernard Hospital
Locations (1):
- AP-HP, Bichat-Claude Bernard Hospital, Paris, France

REFERENCES:
- [Background] Peled Y, Ram E, Lavee J, Sternik L, Segev A, Wieder-Finesod A, Mandelboim M, Indenbaum V, Levy I, Raanani E, Lustig Y, Rahav G. BNT162b2 vaccination in heart transplant recipients: Clinical experience and antibody response. J Heart Lung Transplant. 2021 Aug;40(8):759-762. doi: 10.1016/j.healun.2021.04.003. Epub 2021 Apr 21. PMID 34034958
- [Background] Itzhaki Ben Zadok O, Shaul AA, Ben-Avraham B, Yaari V, Ben Zvi H, Shostak Y, Pertzov B, Eliakim-Raz N, Abed G, Abuhazira M, Barac YD, Mats I, Kramer MR, Aravot D, Kornowski R, Ben-Gal T. Immunogenicity of the BNT162b2 mRNA vaccine in heart transplant recipients - a prospective cohort study. Eur J Heart Fail. 2021 Sep;23(9):1555-1559. doi: 10.1002/ejhf.2199. Epub 2021 May 14. PMID 33963635